CLINICAL TRIAL: NCT07137286
Title: Genetic Influence on LDL Hyper-responsiveness in Patients Following a Ketogenic Diet
Brief Title: A Study of Genetic Influence on LDL Hyper-responsiveness in Patients Following a Ketogenic Diet
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen L. Kopecky, Principal Investigator, Mayo Clinic
Other Study IDs: 25-002523
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: LDL Hyper-responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify whether individuals following a ketogenic diet who experience extreme LDL-C elevation, termed "hyper-responders", have identifiable genetic variations in genes involved in cholesterol absorption.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* LDL-C >170 mg/dL in response to starting a ketogenic diet

Exclusion Criteria:

* Patients who do not consent to blood draw for genetic testing
* Those with LDL-C <170 mg/dL on a ketogenic diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Patients to have a genetic mutation | Baseline
  Genetic Mutation will be defined as a mutation in ABCG5, ABCG8, APOB, APOE, CETP, CYP27A1, LDLR, LDLRAP1, LIPA, LPL, LRP6, and PCSK9 genes

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kopecky, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No